CLINICAL TRIAL: NCT07390097
Title: Effect of Perioperative Calcium Dobesilate on Postprocedural Pain, Symptom Relief, and Quality of Life After Radiofrequency Ablation for Great Saphenous Vein Insufficiency: A Randomized Controlled Trial
Brief Title: Calcium Dobesilate After Radiofrequency Ablation for Varicose Veins
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oguz Arslanturk (Other)
Responsible Party: Sponsor-Investigator, Oguz Arslanturk, Assistant Professor, Department of Cardiovascular Surgery, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BEUN-CVS-2026-001
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Varicose Veins Leg; Great Saphenous Vein Insufficiency; Chronic Venous Insufficiency
Keywords: Calcium Dobesilate; Radiofrequency Ablation; Venoactive Drug; Postoperative Pain; Quality of Life
MeSH Terms: conditions — Pain, Postoperative | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to intervention (calcium dobesilate) or control (standard care) group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants receive standard care only (RFA plus compression stockings) without calcium dobesilate.
- Calcium Dobesilate Group (Experimental): Participants receive calcium dobesilate 500 mg orally twice daily, starting 7 days before RFA and continuing for 30 days after the procedure, in addition to standard care (RFA plus compression stockings).
  Interventions: Drug: calcium dobesilate

INTERVENTIONS:
Drug: calcium dobesilate — Calcium dobesilate 500 mg oral tablet, twice daily (morning and evening), starting 7 days before radiofrequency ablation and continuing for 30 days postoperatively. Total treatment duration is 37 days.
  Arms: Calcium Dobesilate Group

SUMMARY:
This study evaluates whether calcium dobesilate, a venoactive drug, improves recovery after radiofrequency ablation (RFA) for varicose veins. Patients with great saphenous vein insufficiency undergoing RFA will be randomly assigned to receive either calcium dobesilate (500 mg twice daily) or standard care alone. The treatment starts 7 days before the procedure and continues for 30 days after. The primary outcome is postoperative pain at day 7. Secondary outcomes include pain at days 14 and 30, quality of life, ecchymosis, and return to daily activities.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) is a minimally invasive treatment for great saphenous vein insufficiency. Although effective, patients may experience postprocedural pain, ecchymosis, and discomfort during recovery. Venoactive drugs have been shown to reduce symptoms in chronic venous disease and may improve recovery after venous procedures.

Calcium dobesilate is a venoactive agent that reduces capillary permeability, inhibits platelet aggregation, and has anti-inflammatory properties. It is approved for chronic venous insufficiency treatment in many countries including Turkey.

This prospective, randomized, open-label, controlled trial will investigate whether perioperative calcium dobesilate administration improves clinical outcomes after RFA. Approximately 100 patients will be enrolled and randomized 1:1 to either:

* Intervention group: Calcium dobesilate 500 mg twice daily starting 7 days before RFA and continuing for 30 days postoperatively, plus standard care
* Control group: Standard care alone (RFA plus compression stockings)

All patients will undergo standardized RFA procedure under tumescent anesthesia. Assessments will be performed at baseline, and postoperative days 1, 7, 14, 30, and 90. Primary endpoint is pain score (VAS) at day 7. Secondary endpoints include VCSS, CIVIQ-20 quality of life score, ecchymosis score, analgesic use, and time to return to normal activities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Symptomatic primary varicose veins (CEAP classification C2-C4)
* Great saphenous vein insufficiency confirmed by duplex ultrasound (reflux >0.5 seconds)
* Great saphenous vein diameter 5-12 mm
* Scheduled for radiofrequency ablation
* Able to provide written informed consent

Exclusion Criteria:

* History of deep vein thrombosis
* Peripheral arterial disease (ABI <0.9)
* Active venous ulcer (CEAP C6)
* Pregnancy or breastfeeding
* Severe renal or hepatic insufficiency
* Known allergy to calcium dobesilate
* Use of venoactive drugs within the past 4 weeks
* Current anticoagulant therapy
* Previous venous intervention on the same limb
* Bilateral disease requiring simultaneous treatment
* Inability to comply with follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS) | Postoperative day 7
  Pain intensity measured using Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Postoperative Pain Score at Day 14 and Day 30 | Postoperative day 14 and day 30
  Pain intensity measured using Visual Analog Scale (VAS) ranging from 0 to 10
Venous Clinical Severity Score (VCSS) | Baseline, day 30, and day 90
  Clinical assessment of venous disease severity using standardized VCSS scoring system (0-30 points)
Quality of Life (CIVIQ-20) | Baseline, day 14, day 30, and day 90
  Disease-specific quality of life measured using Chronic Venous Insufficiency Questionnaire (CIVIQ-20)
Ecchymosis Score | Postoperative day 1, day 7, and day 14
  Postoperative bruising assessed using a 5-point scale (0=none, 1=<5cm, 2=5-10cm, 3=10-20cm, 4=>20cm)
Time to Return to Normal Activities | Up to 30 days postoperatively
  Number of days until patient returns to normal daily activities and work
Postoperative Paresthesia Incidence | Postoperative day 7, day 30, and day 90
  Presence and severity of numbness, tingling, or sensory changes along the treated vein assessed using a 4-point scale (0=none, 1=mild, 2=moderate, 3=severe)
Endovenous Heat-Induced Thrombosis (EHIT) Incidence | Postoperative day 7
  Presence and grade of thrombus extension into the deep venous system assessed by duplex ultrasound using Lawrence classification (Class 1-4)
Great Saphenous Vein Occlusion Rate | Postoperative day 30 and day 90
  Complete occlusion of treated great saphenous vein confirmed by duplex ultrasound (absence of flow and compressibility)

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Arslanturk, MD, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University Hospital, Department of Cardiovascular Surgery, Kozlu, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to local data protection regulations and limited resources for data anonymization and management.